CLINICAL TRIAL: NCT00799357
Title: Utility of Bedside Ultrasound in the Prediction of Difficult Airway
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Collaborators: The Association for Medical Ultrasound (Other)
Responsible Party: Sponsor
Other Study IDs: 0526-08-EP
Record Dates: First submitted 2008-11-26; First posted 2008-11-27 (Estimated); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Laryngoscopy
Keywords: ultrasound

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess the utility of bedside ultrasound to predict difficult airway in patients requiring emergency intubation.

DETAILED DESCRIPTION:
A variety of pre-intubation clinical screening tests have been advocated to predict difficult laryngoscopy, but their usefulness is limited in emergency department, intensive care unit, pre-hospital and combat settings. Patients in these settings are often confused, lethargic, obtunded, uncooperative and common screening tests for difficult laryngoscopy cannot be applied in a large number of emergency intubations. In the recent past, there has been growing interest in upper airway ultrasound. The purpose of this study is to assess the utility of bedside ultrasound to predict difficult airway in patients requiring emergency intubation.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for any surgery under general anesthesia with endotracheal intubation

Exclusion Criteria:

* Upper airway pathologies (facial fractures, tumours, etc)
* Cervical spine fractures
* Tracheostomy tube
* unable to give consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pre-op patients
Sampling Method: Probability Sample
Enrollment: 162 (Estimated)
Dates: Start 2008-12-09 (Actual); Primary Completion 2009-06-01 (Actual); Study Completion 2009-06-01 (Actual)

PRIMARY OUTCOMES:
Predictors of difficult laryngoscopy | one day

CONTACTS AND LOCATIONS:
Overall Officials: Srikar R Adhikari, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

REFERENCES:
- [Result] Komatsu R, Sengupta P, Wadhwa A, Akca O, Sessler DI, Ezri T, Lenhardt R. Ultrasound quantification of anterior soft tissue thickness fails to predict difficult laryngoscopy in obese patients. Anaesth Intensive Care. 2007 Feb;35(1):32-7. doi: 10.1177/0310057X0703500104. PMID 17323663
- [Result] Ezri T, Gewurtz G, Sessler DI, Medalion B, Szmuk P, Hagberg C, Susmallian S. Prediction of difficult laryngoscopy in obese patients by ultrasound quantification of anterior neck soft tissue. Anaesthesia. 2003 Nov;58(11):1111-4. doi: 10.1046/j.1365-2044.2003.03412.x. PMID 14616599
- [Result] Chou HC, Wu TL. Large hypopharyngeal tongue: a shared anatomic abnormality for difficult mask ventilation, difficult intubation, and obstructive sleep apnea? Anesthesiology. 2001 May;94(5):936-7. doi: 10.1097/00000542-200105000-00043. No abstract available. PMID 11388555